CLINICAL TRIAL: NCT04549805
Title: Troponin Within the Normal Reference Range to Risk Stratify Patients With Acute Chest Pain for Computed Tomography Coronary Angiography
Brief Title: Troponin to Risk Stratify Patients for Computed Tomography Coronary Angiography
Acronym: PRECISE-CTCA
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 245971
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Coronary artery disease; CT coronary angiography; High-sensitivity cardiac troponin
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The study aims to take four blood samples from study participants at time of consent if this is done in person and also at time of CTCA in the intervention arm for long-term storage. The sample types and volumes are detailed below:
  * Plasma Li-Hep (approx. 4.7ml)
  * Serum Gel (approx. 9ml)
  * EDTA (approx. 4.9ml)
  * EDTA (approx. 9ml) Where possible, surplus serum and/or plasma will also be obtained from the clinical blood samples sent by the clinical care team during the initial hospital attendance.
  All samples will be centrifuged and stored at -80 degrees Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients without myocardial injury: Patients without myocardial injury will be recruited in a 2:1 fashion stratified by peak high-sensitivity cardiac troponin I concentration above and below a threshold of 5 ng/L.
  Interventions: Diagnostic Test: Computed Tomography Coronary Angiography

INTERVENTIONS:
Diagnostic Test: Computed Tomography Coronary Angiography — In order to optimise the quality of the Computed Tomography Coronary Angiography scan images, participants might be given tablets or an injection (e.g. beta-blockers, calcium channel antagonist, ivabradine) to slow their heart rate and glyceryl trinitrate (GTN) following local protocol guidance.

SUMMARY:
Most patients presenting to hospital with chest pain are discharged home without further tests once a heart attack has been ruled out. Current strategies to assess patients with a suspected heart attack involve blood tests to measure troponin, a protein released into the bloodstream when the heart muscle is damaged. Despite having had a heart attack ruled-out, some patients have unrecognised coronary heart disease and are at risk of having a heart attack in the future. However, we do not know what is the best approach to identify and treat these patients.

This study will use a heart scan known as computed tomography coronary angiogram (CTCA) to look for underlying coronary heart disease in patients who have had a heart attack ruled out. In an earlier study, we performed this scan in patients referred to the outpatient cardiology clinic with stable chest pain and found that this improved the diagnosis of coronary heart disease, leading to improvement in patient care that prevented many future heart attacks. Our research has also demonstrated that troponin levels below the threshold used to diagnose a heart attack identify those who are at greater risk of having a heart attack in the future. The aim of this study is to confirm whether these low levels of troponin can identify patients who have underlying coronary heart disease and may benefit from further testing and preventative treatment.

DETAILED DESCRIPTION:
Using a newer, more sensitive troponin test, we now know that troponin levels even below the threshold used to diagnose a heart attack identify patients who are at risk of having a heart attack in the future. Our research in patients with stable chest pain demonstrated that computed tomography coronary angiogram (CTCA) improved the diagnosis of coronary heart disease, leading to improvement in patient care that prevented many future heart attacks. This study will build on these two major strands of research to confirm whether these low levels of troponin can identify patients who have underlying coronary heart disease and may benefit from further testing and preventative treatment.

The investigators will evaluate consecutive patients presenting to hospital with suspected acute coronary syndrome and cardiac troponin concentration within the normal reference range for the presence of underlying coronary artery disease. All participants will be invited for an outpatient CTCA.

Findings from this study will help inform a randomised controlled trial to evaluate the role of CTCA in patients who have a heart attack ruled out, but are identified as intermediate risk on troponin testing.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to hospital with acute chest pain or equivalent symptoms of suspected acute coronary syndrome
* Maximum high-sensitivity cardiac troponin I concentration below the 99th centile (16 ng/L for women and 34 ng/L in men)

Exclusion Criteria:

* Diagnosis of myocardial infarction during index presentation
* Clear alternative diagnosis for index presentation
* Recent CT or invasive coronary angiogram (within 1 year)
* Patient inability to undergo CT scanning, due to severe renal failure (estimated glomerular filtration rate <30 mL/min) or major allergy to iodinated contrast media
* Pregnancy or breast feeding
* Inability to give informed consent
* Further investigation for coronary artery disease would not in the patient's interest, due to limited life expectancy, quality of life or functional status

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (30 years and over) with acute chest pain or equivalent symptoms of suspected acute coronary syndrome and maximum high-sensitivity cardiac troponin I concentration below the 99th centile (16 ng/L for women and 34 ng/L in men)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with obstructive coronary artery disease | Ideally within 4 weeks of index presentation
  Proportion of participants with >50% stenosis in the left main stem or >70% stenosis in other coronary arteries

SECONDARY OUTCOMES:
Proportion of participants with moderate non-obstructive coronary artery disease | Ideally within 4 weeks of index presentation
  Proportion of participants with 50-70% stenosis in one or more coronary arteries
Proportion of participants with mild non-obstructive coronary artery disease | Ideally within 4 weeks of index presentation
  Proportion of participants with 10-50% stenosis in one or more coronary arteries
Proportion of participants with insignificant coronary artery disease | Ideally within 4 weeks of index presentation
  Proportion of participants with 1-10% stenosis in one or more coronary arteries
Proportion of participants with normal coronary arteries | Ideally within 4 weeks of index presentation
  Proportion of participants with no stenosis in coronary arteries

OTHER OUTCOMES:
Leaman score for overall coronary artery disease burden | Ideally within 4 weeks of index presentation
Proportion of participants with adverse coronary artery plaque features | Ideally within 4 weeks of index presentation
Myocardial mass | Ideally within 4 weeks of index presentation
Proportion of participants with hemodynamically significant coronary stenosis on CT-derived fractional flow reserve (CT-FFR) | Ideally within 4 weeks of index presentation
Left ventricular volume | Ideally within 4 weeks of index presentation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Requests for IPD will be considered on an individual basis.

REFERENCES:
- [Derived] Perez-Vicencio D, Thurston AJF, Doudesis D, O'Brien R, Ferry A, Fujisawa T, Williams MC, Gray AJ, Mills NL, Lee KK. Risk scores and coronary artery disease in patients with suspected acute coronary syndrome and intermediate cardiac troponin concentrations. Open Heart. 2024 Aug 3;11(2):e002755. doi: 10.1136/openhrt-2024-002755. PMID 39097328